CLINICAL TRIAL: NCT01360866
Title: A Long-term, Phase 3, Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Oral OPC-34712 as Adjunctive Therapy in Adults With Major Depressive Disorder, the Orion Trial
Brief Title: Safety and Tolerability of Oral OPC-34712 as Adjunctive Therapy in Adults With Major Depressive Disorder (the Orion Trial)
Acronym: Orion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-10-238
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders
Keywords: OPC-34712; brexpiprazole; Major Depressive Disorder; Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders | interventions — Escitalopram; Fluoxetine; Paroxetine; Sertraline; Duloxetine Hydrochloride; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- OPC-34712 (Brexpiprazole) and Escitalopram (Experimental): OPC-34712: Oral tablet; 0.5 to 3 mg/day Escitalopram: Oral tablet; 10 or 20 mg/day
  Interventions: Drug: OPC-34712; Drug: Escitalopram
- OPC-34712 and Fluoxetine (Experimental): OPC-34712: Oral tablet; 0.5 to 3 mg/day Fluoxetine: Oral capsules; 20 or 40 mg/day
  Interventions: Drug: OPC-34712; Drug: Fluoxetine
- OPC-34712 and Paroxetine CR (Experimental): OPC-34712: Oral tablet; 0.5 to 3 mg/day Paroxetine CR: Oral controlled-release tablets; 37.5 or 50 mg/day
  Interventions: Drug: OPC-34712; Drug: Paroxetine CR
- OPC-34712 and Sertraline (Experimental): OPC-34712: Oral tablet; 0.5 to 3 mg/day Sertraline: Oral tablets; 100, 150, or 200 mg/day
  Interventions: Drug: OPC-34712; Drug: Sertraline
- OPC-34712 and Duloxetine (Experimental): OPC-34712: Oral tablet; 0.5 to 3 mg/day Duloxetine: Oral delayed-release capsules; 40 or 60 mg/day
  Interventions: Drug: OPC-34712; Drug: Duloxetine
- OPC-34712 and Venlafaxine XR (Experimental): OPC-34712: Oral tablet; 0.5 to 3 mg/day Venlafaxine XR: Oral extended-release capsules; 75, 150, or 225 mg/day
  Interventions: Drug: OPC-34712; Drug: Venlafaxine XR

INTERVENTIONS:
Drug: OPC-34712 — Tablet
Drug: Escitalopram — Tablet
  Other Names: Lexapro
  Arms: OPC-34712 (Brexpiprazole) and Escitalopram
Drug: Fluoxetine — Capsule
  Other Names: Prozac
  Arms: OPC-34712 and Fluoxetine
Drug: Paroxetine CR — Controlled-release tablets
  Other Names: Paxil CR
  Arms: OPC-34712 and Paroxetine CR
Drug: Sertraline — Tablets
  Other Names: Zoloft
  Arms: OPC-34712 and Sertraline
Drug: Duloxetine — Delayed-release capsules
  Other Names: Cymbalta
  Arms: OPC-34712 and Duloxetine
Drug: Venlafaxine XR — Extended-release capsules
  Other Names: Effexor XR
  Arms: OPC-34712 and Venlafaxine XR

SUMMARY:
To assess the long-term safety and tolerability of oral OPC-34712 (brexpiprazole), given in addition to an FDA approved antidepressant (ADT) for the treatment of adults with Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Male and Female outpatients 18-65 years of age

Eligible subjects from Trials 331-10-227, 331-10-228 or 331-12-282:

* Subjects who completed participation in the Double-blind Randomization Phase (i.e. Week 14 visit) in Trial 331-10-227, Trial 331-10-228, or Trial 331-12-282 or
* Subjects who met criteria for a response, but did not meet criteria for remission at Week 14 of either trial

Eligible subjects from other Phase 3, Double-blind, Brexpiprazole MDD trials:

• Subjects who completed the last scheduled visit of the prior Double-blind Randomized Phase 3 trial.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving OPC-34712.
* Subjects with a major protocol violation during the course of their participation in the Double-blind Randomization Phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2944 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (142):
- United States (93):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Costa Mesa, California
  - Research Site, Glendale, California
  - Research Site, Irvine, California
  - Research Site, Oceanside, California
  - Research Site, Redlands, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Ana, California
  - Research Site, Sherman Oaks, California
  - Research Site, Temecula, California
  - Research Site, Upland, California
  - Research Site, Norwalk, Connecticut
  - Research Site, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Oakland Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, The Villages, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Oak Brook, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lake Charles, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Belmont, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Methuen, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Weymouth, Massachusetts
  - Research Site, Rochester Hills, Michigan
  - Research Site, Creve Coeur, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Tom River, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Jamaica, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Bridgeville, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Lincoln, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Murray, Utah
  - Research Site, Woodstock, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Herndon, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Brown Deer, Wisconsin
  - Research Site, Middleton, Wisconsin
- Canada (5):
  - Research Site, Gatineau
  - Research Site, Penticton
  - Research Site, Pointe-Claire
  - Research Site, Sherbrooke
  - Research Site, Toronto
- France (7):
  - Research Site, Arcachon
  - Research Site, Douai
  - Research Site, Élancourt
  - Research Site, Jarnac
  - Research Site, Orvault
  - Research Site, Palaiseau
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Achim
  - Research Site, Bochum
  - Research Site, Mittweida
  - Research Site, Stralsund
  - Research Site, Würzburg
- Research Site, Budapest, Hungary
- Poland (9):
  - Research Site, Bełchatów
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Pruszcz Gdański
  - Research Site, Tuszyn
  - Research Site, Wroclaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Târgu Mureş
- Russia (8):
  - Research Site, Arkhangelsk Region
  - Research Site, Moscow
  - Research Site, Roshchino
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersberg
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Tonnel’nyy
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Kneževac
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Michalovce
- Ukraine (4):
  - Research Site, Chernihiv
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Poltava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newcomer JW, Meehan SR, Chen D, Brubaker M, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Prediabetes Treated With Adjunctive Brexpiprazole for Major Depressive Disorder: Pooled Analysis of Short- and Long-Term Clinical Studies. J Clin Psychiatry. 2023 Aug 28;84(5):23m14786. doi: 10.4088/JCP.23m14786. PMID 37656180
- [Derived] Newcomer JW, Eriksson H, Zhang P, Meehan SR, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Major Depressive Disorder Treated With Adjunctive Brexpiprazole: Pooled Analysis of Phase 3 Clinical Studies. J Clin Psychiatry. 2019 Oct 1;80(6):18m12680. doi: 10.4088/JCP.18m12680. PMID 31577867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 2944 participants at 188 sites in 11 countries: Canada, France, Germany, Hungary, Poland, Romania, Russian Federation, Serbia, Slovakia, Ukraine, and United States (US).
Pre-assignment Details: The study population consisted of eligible participants who completed one of the double-blind, phase 3 brexpiprazole major depressive disorder (MDD) trials and who, could potentially benefit from adjunctive treatment with oral brexpiprazole for MDD.
Groups:
- Prior Placebo: Participants who received placebo with antidepressant therapy [ADT] in previous double blind phase 3 studies, received 0.5 to 3 mg/day Brexpiprazole + ADT for weeks 1, 2, 4, 8,14, 20, 26, 32, 38, 44 and 52 with dose adjustment.
- Prior Brexpiprazole: Participants who received Brexpiprazole with ADT in previous double blind phase 3 studies, received 0.5 to 3 mg/day Brexpiprazole + ADT for weeks 1, 2, 4, 8,14, 20, 26, 32, 38, 44 and 52 with dose adjustment.
- Prior ADT: Participants who received only ADT in previous double blind phase 3 studies and were not randomized, received 0.5 to 3 mg/day Brexpiprazole + ADT for weeks 1, 2, 4, 8,14, 20, 26, 32, 38, 44 and 52 with dose adjustment.
- Prior Seroquel: Participants who received Seroquel with ADT in previous double blind phase 3 studies, received 0.5 to 3 mg/day Brexpiprazole + ADT for weeks 1, 2, 4, 8,14, 20, 26, 32, 38, 44 and 52 with dose adjustment.
Period: Overall Study
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
Started | 516 | 707 | 1645 | 76
Completed | 295 | 420 | 1126 | 54
Not Completed | 221 | 287 | 519 | 22
Not completed — Lost to Follow-up | 11 | 28 | 41 | 0
Not completed — Adverse Event | 56 | 61 | 134 | 6
Not completed — Paticipant met withdrawal criteria | 11 | 28 | 54 | 0
Not completed — Withdrawn by Investigator | 9 | 8 | 31 | 2
Not completed — Withdrawal by participant | 79 | 89 | 168 | 8
Not completed — Protocol Deviation | 25 | 33 | 61 | 2
Not completed — Lack of Efficacy | 30 | 40 | 30 | 4

BASELINE CHARACTERISTICS:
Population: comprised of all participants who signed an informed consent form (ICF) for the trial.
Groups:
- Prior Placebo: Participants who received placebo with ADT in previous double blind phase 3 studies, received 0.5 to 3 mg/day Brexpiprazole + ADT for weeks 1, 2, 4, 8,14, 20, 26, 32, 38, 44 and 52 with dose adjustment.
- Prior ADT: Participants who received only ADT in previous double blind phase 3 studies, received 0.5 to 3 mg/day Brexpiprazole + ADT for weeks 1, 2, 4, 8,14, 20, 26, 32, 38, 44 and 52 with dose adjustment.
- Total: Total of all reporting groups
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel | Total
Number analyzed (Participants) | 516 | 707 | 1645 | 76 | 2944
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (11.0) | 45.0 (11.0) | 44.0 (12.0) | 44.0 (11.0) | 45.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367 | 479 | 1108 | 51 | 2005
  Male | 149 | 228 | 537 | 25 | 939
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 452 | 609 | 1459 | 68 | 2588
  Black or African American | 55 | 76 | 149 | 8 | 288
  American Indian or Alaska Native | 0 | 6 | 8 | 0 | 14
  Asian | 5 | 8 | 8 | 0 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 6 | 0 | 6
  Other | 4 | 8 | 15 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) - All Participants
Description: To assess the frequency and severity of AEs as the variables of safety and tolerability of brexpiprazole.
Time Frame: From screening to week 52/early termination
Population: Participants who received at least one dose of open-label brexpiprazole as adjunctive therapy to one of the allowed ADTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
Number analyzed (Participants) | 516 | 706 | 1640 | 76
Participants
  Participants with adverse events | 400 | 511 | 1165 | 51
  Participants with treatment emergent AE (TEAE) | 399 | 510 | 1163 | 51
  Participants with serious TEAE | 14 | 23 | 33 | 1
  Participants with severe TEAE | 48 | 64 | 99 | 4
  Partcipants discontinued due to AEs | 55 | 58 | 134 | 6

2. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression - Severity (CGI-S) of Illness Score
Description: The severity of illness for each participant was rated using the CGI-S . On the basis of the investigator answer to the question: "Considering your total clinical experience with this particular population, how mentally ill was the participant at that time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: From screening to week 52/early termination
Population: Participants who received at least one dose of open-label brexpiprazole as adjunctive therapy to one of the allowed ADTs and had at least one post-baseline efficacy evaluation of CGI-S.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
Number analyzed (Participants) | 512 | 698 | 1630 | 76
units on a scale | -0.77 (1.11) | -0.63 (1.16) | -0.48 (1.04) | -0.93 (0.85)

3. Secondary Outcome: Change From Baseline in Mean Clinical Global Impression - Improvement (CGI-I) Score
Description: The efficacy of trial treatment was rated for each participant using the CGI-I. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. All responses were compared to the participant's condition at screening. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse and 7 = very much worse.
Time Frame: From screening to week 52/early termination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
Number analyzed (Participants) | 505 | 693 | 1606 | 75
units on a scale | 2.60 (1.30) | 2.63 (1.34) | 2.63 (1.39) | 2.40 (1.17)

4. Secondary Outcome: Summary of Mean Change From Baseline in Sheehan Disability Scale (SDS) Mean Score
Description: The SDS was a self-rated instrument used to measure the effect of the participant's symptoms on regular life responsibilities. The SDS was a visual analogue scale that used spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the 3 domains with scores from 0 = not at all, to 10 = extremely.
  Scores of 5 and above were associated with significant functional impairment.
Time Frame: From screening to week 52/early termination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
Number analyzed (Participants) | 346 | 457 | 1165 | 53
units on a scale | -0.80 (2.80) | -0.70 (2.60) | -0.40 (2.30) | -1.00 (1.70)

5. Secondary Outcome: Change From Baseline in the Inventory of Depressive Symptomatology - Self Report (IDS-SR) Total Score
Description: The IDS-SR was a 30-item self-report measure used to assess core diagnostic depressive symptoms as well as atypical and melancholic symptom features of MDD. The IDS-SR consists of 30 items, all rated on a 0 to 3 scale with 0 being the "best" rating and 3 being the "worst" rating. The IDS-SR Total Score is the sum of ratings of 28 item scores. The possible IDS-SR Total Score ranges from 0 (best) to 84 (worst).
  Under item 9, two sub-items 9A and 9B exist, with possible scores of 1, 2 or 3 for item 9A, and 0 or 1 for item 9B. The scores for these two sub-items are not included in the calculation of the total score. Item 11 or item 12 should be completed but not both, and similarly, item 13 or item 14 should be completed but not both. If the number of items recorded is at least 23 and at most 27, the IDS-SR Total Score will be the mean of the recorded items multiplied by 28 and then rounded to the first decimal place.
Time Frame: From screening to week 52/early termination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
Number analyzed (Participants) | 491 | 664 | 1556 | 75
units on a scale | -5.25 (12.21) | -4.76 (11.79) | -3.94 (10.57) | -7.44 (8.89)

ADVERSE EVENTS:
Time Frame: From screening to 30 (+ 2) days following the 52 weeks treatment period or early termination.
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related.
  An AE was considered serious if it resulted in any of the following outcomes: fatal; life threatening; persistently or significantly disabling or incapacitating; required inpatient hospitalization or prolonged existing hospitalization; a congenital anomaly/birth defect; or other medically significant event
Arm/Group | Prior Placebo | Prior Brexpiprazole | Prior ADT | Prior Seroquel
All-Cause Mortality (participants affected / at risk) | 2/516 | 2/706 | 0/1640 | 0/76
Serious Adverse Events (participants affected / at risk) | 14/516 | 23/706 | 33/1640 | 1/76
Other Adverse Events (participants affected / at risk) | 296/516 | 323/706 | 787/1640 | 33/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo (N=516) | Prior Brexpiprazole (N=706) | Prior ADT (N=1640) | Prior Seroquel (N=76)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0
Retinal Vein Thrombosis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 2 | 0
Drug Withdrawal Syndrome (General disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Extrapyramidal Disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Ruptured Cerebral Aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Completed Suicide (Psychiatric disorders) | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 2 | 3 | 3 | 0
Depressive Symptom (Psychiatric disorders) | 0 | 0 | 1 | 0
Intentional Self-Injury (Psychiatric disorders) | 0 | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 2 | 1 | 1 | 0
Renal Disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pelvic Adhesions (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic Obstructive Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo (N=516) | Prior Brexpiprazole (N=706) | Prior ADT (N=1640) | Prior Seroquel (N=76)
Constipation (Gastrointestinal disorders) | 14 | 15 | 33 | 4
Nausea (Gastrointestinal disorders) | 26 | 32 | 61 | 4
Fatigue (General disorders) | 37 | 50 | 88 | 3 — General Disorders and Administration Site Conditions
Viral Upper Respiratory Tract Infection (Infections and infestations) | 25 | 35 | 98 | 2
Weight Increased (Investigations) | 118 | 100 | 296 | 5
Increased Appetite (Metabolism and nutrition disorders) | 37 | 28 | 117 | 3
Akathisia (Nervous system disorders) | 54 | 37 | 99 | 7
Headache (Nervous system disorders) | 42 | 55 | 105 | 9
Somnolence (Nervous system disorders) | 40 | 60 | 130 | 5
Anxiety (Psychiatric disorders) | 39 | 37 | 76 | 0
Insomnia (Psychiatric disorders) | 30 | 40 | 108 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

DOCUMENTS (2):
  • Study Protocol (2014-06-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT01360866/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT01360866/SAP_001.pdf